CLINICAL TRIAL: NCT01284946
Title: A Phase II, Open Label Clinical Trial Exploring the Safety and the Efficacy of Oral Deferasirox in Patients Newly Diagnosed With Porphyria Cutanea Tarda (PCT) and Non-transfusion Iron Overload
Brief Title: Safety and Efficacy of Oral Deferasirox in Patients With Porphyria Cutanea Tarda
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Association pour l'Etude des Fonctions Digestives (AEFD) (Unknown)
Responsible Party: COFFIN, Association pour l'Etude des Fonctions Digestives
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AEFD2010-01
Record Dates: First submitted 2011-01-26; First posted 2011-01-27 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2011-01

CONDITIONS: Porphyria Cutanea Tarda
Keywords: PCT sporadic or familial; Skin fragility and bullae lesions; non-transfusion iron overload
MeSH Terms: conditions — Porphyria Cutanea Tarda | interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exjade (Experimental): Safety and efficacy
  Interventions: Drug: Exjade

INTERVENTIONS:
Drug: Exjade — Orodispersible Tablet, 10 mg/Kg/day ± 5 mg/Kg/day during 24 weeks Deferasirox should be taken daily 30 minutes before breakfast
  Other Names: DEFERASIROX

SUMMARY:
While clinical phlebotomy is current standard practice for alleviating non-transfusion iron overload in patients with PCT, it may not be suitable for all patients. For example, some patients are unwilling to be adequately phlebotomized because of inconvenience, as phlebotomy can be cumbersome, especially during the induction treatment phase requiring frequent clinic visits (twice a month, for at least 6 months) or because of venous access difficulties. Other patients are unable to undergo phlebotomy due to medical reasons such as anemia or cardiopulmonary disorders. It is postulated such patients with PCT who have non-transfusion iron overload could benefit from treatment with deferasirox (Exjade®), a once daily oral iron chelator licensed in several countries, including the EU, for treating transfusion iron overload in adult and pediatric patients. Although there is some data on the efficacy and safety of deferasirox in patients with HH, who, like those with PCT, have non-transfusional iron overload, there is a need to evaluate the safety and efficacy of deferasirox treatment of non-transfusion iron overload in patients with PCT.

DETAILED DESCRIPTION:
The primary objective is to assess the safety of deferasirox in treating non-transfusion iron overload in patients with PCT.

The secondary objective is to assess the effectiveness of deferasirox treatment :

After 3 and 6 months to:

•Lower serum ferritin from abnormal to normal standard ranges specified for males and females in this patient population.

After 6 months to :

•Lower liver iron content after 24 weeks of treatment measured by liver MRI T2

After 3 and 6 months to :

* Improve clinical symptoms, i.e. improvement in skin lesions (reduction or no new bullae formation), and skin fragility (photographs will be used).
* Reduce porphyrin levels.

ELIGIBILITY:
Inclusion Criteria:

* Male and female diagnosed with clinically overt Porphyria Cutanea Tarda, sporadic or familial as per the European Porphyria Network guidelines i.e. increased urinary and plasma porphyrins and faecal isocoproporphyrin detected by fluorescence emission spectroscopy,

  * Skin fragility and bullae lesions,
  * Age ≥ 18 years old,
  * non-transfusion iron overload as depicted by a serum ferritin value ≥ 300 μg/L for men and ≥ 200 μg/L for women, and/or LIC ≥ 2 mg Fe/g dw for both men and women and with transferrin saturation ≥ 45%,
  * Adequate liver function i.e. ALAT/ASAT and Alkaline Phosphatase ? 2.5 times ULN, bilirubin < 1.5 times ULN,
  * Signed informed consent prior to beginning the specific procedures of the protocol,
  * Ability to comply with all study-related procedures, medications, and evaluations,
  * Sexually active women must use an effective method of contraception, or must have undergone clinically documented total hysterectomy and/or oophorectomy, or tubal ligation or be postmenopausal (defined as amenorrhea for at least 12 months). Since hormonal therapy may cause PCT, oral contraceptives will not be started during the course of the study and patients already on oral contraceptives will be advised to speak to their physician about discontinuing them and will not be enrolled in the study.

Exclusion Criteria:

* Clinical evidence of active Hepatitis B (positive HBsAg with negative HBsAb) and/or hepatitis C (positive HCV antibody and detectable HCV RNA with ALT above the normal range)

  * Patients with on going alcoholic dependency > 60g/day
  * Serum creatinine above the ULN
  * Creatinine clearance < 60 ml/min, estimated according to Cockcroft-Gault formula or MDRD formula for adults
  * Significant proteinuria as indicated by a urine protein: urine creatinine ratio > 0.5 mg/mg in a non-first void urine sample.
  * Diabetes
  * Iron overload due to hereditary hemochromatosis
  * History of blood transfusion during the 6 months prior to study entry,
  * Males with hemoglobin <13 mg/dL, females with hemoglobin <12 mg/dL
  * Active peptic ulcus
  * Treatment with phlebotomy within 2 weeks of screening visit
  * Prior Desferal® treatment within 1 month of the screening visit
  * Patients currently or previously treated with deferiprone or deferasirox
  * Patients with a diagnosis of a clinically relevant cataract or a previous history of clinically relevant ocular toxicity related to iron chelation
  * Patient with clinically significant decrease of hearing
  * Pregnant or lactating women or women of childbearing potential not using adequate contraception (pregnancy test mandatory and negative for patient with childbearing potential)
  * Known hypersensitivity to the active ingredient of deferasirox or any excipients
  * Contraindication to the administration of deferasirox as outlined in the approved prescribing information.
  * Presence of a surgical or medical condition that might significantly alter the absorption, distribution, metabolism or excretion of deferasirox
  * Presence of a non-controlled severe disease affected vital organs as cardiac and/or pulmonary disease
  * Patients with a known diagnosis of cirrhosis (confirmed by biopsy)
  * Patients with active inflammatory diseases that may interfere with the accurate measurement of serum ferritin
  * Patients treated with systemic investigational drug within 4 weeks prior or with topical investigational drug within 7 days prior to the screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to assess the safety of deferasirox in treating non-transfusion iron overload in patients with PCT. | 6 months
Related drug adverse events | 6 months
  Incidence type and severity of drug related adverse events

SECONDARY OUTCOMES:
The change from baseline in serum ferritin after 12 and 24 weeks of treatment,The change from baseline in iron burden after 24 weeks of treatment measured by liver MRI T2,The evolution of clinical symptoms | 6 months
Chage from baseline in serum ferritin, iron burden, improvement in clincal symptoms, porphyrin levels | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Deybach Jean-Charles, Professor, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Louis Mourier, GI unit,, Colombes, Île-de-France Region, France

REFERENCES:
- [Result] Puy H, Gouya L, Deybach JC. Porphyrias. Lancet. 2010 Mar 13;375(9718):924-37. doi: 10.1016/S0140-6736(09)61925-5. PMID 20226990